CLINICAL TRIAL: NCT01045148
Title: Virtual HDR CyberKnife Radiosurgery for Localized Prostatic Carcinoma: A Phase II Study
Brief Title: CyberKnife Radiosurgery for Localized Prostatic Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CyberKnife Centers of San Diego (Other)
Responsible Party: Principal Investigator, Carlyn Tripp, Donald Fuller, M.D., CyberKnife Centers of San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Virtual HDR CK Radiosurgery
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
Keywords: Prostatic Cancer; Prostatic Neoplasms; Prostate Neoplasms; Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CyberKnife Radiosurgery (Other): CyberKnife Radiosurgery
  Interventions: Radiation: CyberKnife Radiosurgery

INTERVENTIONS:
Radiation: CyberKnife Radiosurgery — High Dose 3800 cGy/4 fractions
Radiation: CyberKnife Radiosurgery — Moderate Dose 3400 cGy/5 fractions

SUMMARY:
Virtual high dose rate (HDR) CyberKnife (CK) prostate treatment has comparable morbidity and efficacy compared with actual prostate HDR treatment, but does it without the catheters and hospital admission. As such, it is a more "patient friendly" treatment method compared with actual prostate HDR brachytherapy as currently practiced. Related, as has previously been reported with actual prostate HDR treatment, Virtual HDR CyberKnife prostate treatment should have a high efficacy but with lower acute and chronic morbidity compared with other local prostate cancer treatment methods such as permanent seed prostate brachytherapy.

DETAILED DESCRIPTION:
Brachytherapy is a form of treatment where a radioactive isotope is implanted directly into a tumor volume to deliver a lethal dose of radiation. High Dose Rate (HDR) Prostate brachytherapy is a particularly elegant brachytherapy dose sculpting method that is effectively used in the curative treatment of prostate cancer; however, it requires hospital admission and many temporarily implanted transperineal catheters to deliver the radiation source to the target volume, resulting in significant patient discomfort. CyberKnife delivers a form of radiation treatment that is so precise, it appears capable of reconstructing HDR prostate radiation dose sculpting, without the hospital admission and without the catheters. The CyberKnife device is also used for classic radiosurgery, with accuracy comparable to the Gamma Knife, but unlike the Gamma Knife, has the capability to target lesions anywhere in the body with similar accuracy. The aim of this study is to compare CyberKnife morbidity and efficacy with that of HDR and other local treatment methods such a permanent seed prostate brachytherapy in the treatment of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate, clinical stage T1b - T2b (AJCC 6th Edition, see Appendix II), NX/N0, M0.
* Karnofsky performance status > 80.
* Patient must be ≥ 18 years of age.

  * Gleason Sum < or = 7
  * Prostate-specific antigen < or = 20 ng/ml
* Patients must sign a study-specific informed consent form prior to study entry.

Exclusion Criteria:

* Stage < T1b, T2c, T3 or T4 disease (AJCC 6th Edition, see Appendix II).
* Gleason Score > 7.
* PSA > 20 ng/ml.
* Lymph node involvement (N1).
* Evidence of distant metastases (M1).
* Radical surgery for carcinoma of the prostate, prior pelvic radiation, pelvic surgical clips or other metallic foreign bodies.
* History of hormonal therapy (antiandrogen or 5 alpha reductase treatment within three months prior to treatment).
* Previous or concurrent cancers other than basal, in situ, or squamous cell skin cancers unless disease-free for ≥ 5 years.
* Major medical or psychiatric illness, which in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.
* Metallic Hip prosthesis.
* History of inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2006-03; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of CK prostate radiosurgery in terms of morbidity/QOL, relative to other commonly used methods of prostate cancer treatment and the pattern of PSA decline and biochemical relapse-free survival thereafter. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Fuller, M.D., Principal Investigator — CyberKnife Centers of San Diego/Radiation Medical Group- Genesis Healthcare Partners
Locations (1):
- CyberKnife Centers of San Diego, San Diego, California, United States

REFERENCES:
- [Derived] De Bari B, Daidone A, Alongi F. Is high dose rate brachytherapy reliable and effective treatment for prostate cancer patients? A review of the literature. Crit Rev Oncol Hematol. 2015 Jun;94(3):360-70. doi: 10.1016/j.critrevonc.2015.02.003. Epub 2015 Feb 17. PMID 25819287